CLINICAL TRIAL: NCT03301142
Title: Randomized Trial Comparing the Use of Laser and of Kinesiotherapy for the Treatment of Female Stress Urinary Incontinence - a Pilot Study
Brief Title: Study Comparing the Use of Laser and of Kinesiotherapy for the Treatment of Female Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Lucilia Carvalho da Fonseca, Principal investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13341
Record Dates: First submitted 2016-08-10; First posted 2017-10-04 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Urinary Stress Incontinence
Keywords: urinary stress incontinence; urinary incontinence,stress; laser; physiotherapy; kinesiotherapy
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device laser (Experimental): treatment with application of Erbium Laser: YAG 2940nm, SMOOTH mode, one session per month for three months (n=20
  Interventions: Procedure: Laser
- kinesiotherapy (Active Comparator): with supervision twice a week for three months (n=20)
  Interventions: Procedure: kinesiotherapy

INTERVENTIONS:
Procedure: Laser — The patients will be submitted to application of the Erbium Laser: YAG(yttrium aluminium garnet) 2940nm, SMOOTH mode developed by FOTONA.The vaginal canal will be accessed using a specific speculum. The 90 degree laser tip shall be used to perform 4 applications to the anterior and lateral vaginal wall at each of the 5 clock points (9,10:30,12,1:30,3 'o´-clock´), commencing at the back of the vagina, retracting in increments of 0.5cm, where 4 shots are made at each interval up to a distance 1cm short of the external opening of the urethra. After completion of this stage, the 90 degree tip shall be switched for the 360 degree tip, whereupon 4 additional applications shall be performed with 4 shots every 0.5 cm along the vaginal trajectory outlined above.
  Arms: Device laser
Procedure: kinesiotherapy — Patients will be guided by the physiotherapist to perform exercises to strengthen the pelvic floor muscles at home on a daily basis in the supine position with an empty bladder. It will be performed 10 repetitions of five-second contractions, the 15 three-second contractions; 20 two seconds contractions; 20 contractions of a second; 5 repetitions of strong contractions while coughing; 10 repetitions of exercise "bridge" associated with pelvic floor contraction and relaxation up in descending.The level of difficulty in performing the exercises will be determined in accordance with the adopted position. In .changes position should be held every four sessions.
  Arms: kinesiotherapy

SUMMARY:
The purpose of this study is compare the effect of laser and of kinesiotherapy in the treatment of women with stress urinary incontinence

DETAILED DESCRIPTION:
the objective of this project is to compare the effect of laser and of kinesiotherapy in the treatment of women with stress urinary incontinence. A randomized controlled clinical trial is proposed involving 40 women diagnosed with stress urinary incontinence randomized into two groups: 1) treatment with application of Erbium Laser: YAG 2940nm, SMOOTH mode, one session per month for three months (n=20); 2) treatment with kinesiotherapy for three months with supervision twice a week (n=20). At baseline assessment, patients shall undergo anamnesis, general physical and gynecological exam, assessments of the pelvic floor based on the modified Oxford scale and of the presence of prolapse using the Pelvic Organ Prolapse Quantification (POP-Q) system. The following exams shall also be performed: Type 1 urine, urine culture, urodynamic study and 1-hour Pad test. Participants shall complete both the King's Health Questionnaire and Incontinence Quality of Life Questionnaire (IQOL). Post-treatment, patients will be assessed during follow-up visits at 1, 3, 6 and 12 months by physical exam and application of the questionnaires. The Pad test will be re-administered at 6 and 12 months. Data will be grouped and statistically assessed.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with stress urinary incontinence will be recruited for this study.

Exclusion Criteria:

* Patients presenting detrusor hyperactivity,stress urinary incontinence with sphincter deficiency genital prolapse, stages 3 and 4 on the POP-Q system, genital cancer, history of painful bladder syndrome, previous history of radiotherapy, keloid, use of photosensitive drugs, uncontrolled diabetes mellitus, active vaginal infection (bacterial vaginosis and candidiasis), abnormal genital bleeding or vaginal stenosis shall be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of urinary loss | twelve months
  the urinary loss will be evaluated with the pad test

SECONDARY OUTCOMES:
improvement of pelvic floor strength | twelve months
  Functional evaluation of the pelvic floor with modified Oxford scale

OTHER OUTCOMES:
impact in the quality of life | twelve months
  the impact in the quality of life will be evaluated with the quality of life questionnaires ( King's Health Questionnaire and IQOL quality of life questionnaires).

CONTACTS AND LOCATIONS:
Overall Officials: LUCILIA C FONSECA, Principal Investigator — UNIVERSIDADE SÃO PAULO (USP)
Locations (1):
- Department of Gynecology and Obstetrics of the Clinicas Hospital of the (FMUSP)., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrams P, Blaivas JG, Stanton SL, Andersen JT. The standardisation of terminology of lower urinary tract function. The International Continence Society Committee on Standardisation of Terminology. Scand J Urol Nephrol Suppl. 1988;114:5-19. No abstract available. PMID 3201169
- [Result] Subak LL, Brown JS, Kraus SR, Brubaker L, Lin F, Richter HE, Bradley CS, Grady D; Diagnostic Aspects of Incontinence Study Group. The "costs" of urinary incontinence for women. Obstet Gynecol. 2006 Apr;107(4):908-16. doi: 10.1097/01.AOG.0000206213.48334.09. PMID 16582131
- [Result] Rovner ES, Wein AJ. Treatment options for stress urinary incontinence. Rev Urol. 2004;6 Suppl 3(Suppl 3):S29-47. PMID 16985862
- [Result] Herbison GP, Dean N. Weighted vaginal cones for urinary incontinence. Cochrane Database Syst Rev. 2013 Jul 8;2013(7):CD002114. doi: 10.1002/14651858.CD002114.pub2. PMID 23836411
- [Result] Gilpin SA, Gosling JA, Smith AR, Warrell DW. The pathogenesis of genitourinary prolapse and stress incontinence of urine. A histological and histochemical study. Br J Obstet Gynaecol. 1989 Jan;96(1):15-23. doi: 10.1111/j.1471-0528.1989.tb01570.x. PMID 2923839
- [Result] Falconer C, Ekman G, Malmstrom A, Ulmsten U. Decreased collagen synthesis in stress-incontinent women. Obstet Gynecol. 1994 Oct;84(4):583-6. PMID 8090397
- [Result] Konstantinos H, Eleni K, Dimitrios H. Dilemmas in the management of female stress incontinence: the role of pelvic floor muscle training. Int Urol Nephrol. 2006;38(3-4):513-25. doi: 10.1007/s11255-006-0085-3. Epub 2006 Nov 29. PMID 17136582
- [Result] Mouritsen L, Schiotz HA. Pro et contra pelvic floor exercises for female stress urinary incontinence. Acta Obstet Gynecol Scand. 2000 Dec;79(12):1043-5. PMID 11130084
- [Result] Fistonic N, Fistonic I, Gustek SF, Turina IS, Marton I, Vizintin Z, Kazic M, Hreljac I, Perhavec T, Lukac M. Minimally invasive, non-ablative Er:YAG laser treatment of stress urinary incontinence in women--a pilot study. Lasers Med Sci. 2016 May;31(4):635-43. doi: 10.1007/s10103-016-1884-0. Epub 2016 Feb 9. PMID 26861984
- [Result] Posten W, Wrone DA, Dover JS, Arndt KA, Silapunt S, Alam M. Low-level laser therapy for wound healing: mechanism and efficacy. Dermatol Surg. 2005 Mar;31(3):334-40. doi: 10.1111/j.1524-4725.2005.31086. PMID 15841638
- [Result] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Result] Rodrigues AM, de Oliveira LM, Martins Kde F, Del Roy CA, Sartori MG, Girao MJ, Castro Rde A. [Risk factors for genital prolapse in a Brazilian population]. Rev Bras Ginecol Obstet. 2009 Jan;31(1):17-21. doi: 10.1590/s0100-72032009000100004. Portuguese. PMID 19347224
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Result] Tamanini JT, D'Ancona CA, Botega NJ, Rodrigues Netto N Jr. [Validation of the Portuguese version of the King's Health Questionnaire for urinary incontinent women]. Rev Saude Publica. 2003 Apr;37(2):203-11. doi: 10.1590/s0034-89102003000200007. Epub 2003 Apr 4. Portuguese. PMID 12700842
- [Result] Souza CC, Rodrigues AM, Ferreira CE, Fonseca ES, di Bella ZI, Girao MJ, Sartori MG, Castro RA. Portuguese validation of the Urinary Incontinence-Specific Quality-of-Life Instrument: I-QOL. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1183-9. doi: 10.1007/s00192-009-0916-8. Epub 2009 Jun 9. PMID 19506791
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601